CLINICAL TRIAL: NCT03486236
Title: A Phase 1, Randomized, Double Blind, Placebo Controlled, Multiple Dose Escalation Study Evaluating Safety and Pharmacokinetics of VX-440 in Combination With VX-661/Ivacaftor in Healthy Adult Subjects
Brief Title: A Study Evaluating Safety and Pharmacokinetics of VX-440 in Combination With Tezacaftor/Ivacaftor in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX16-440-002; 2016-000762-38 (EudraCT Number)
Record Dates: First submitted 2018-03-27; First posted 2018-04-03 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — tezacaftor; ivacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort C1 (Experimental)
  Interventions: Drug: VX-440; Drug: TEZ; Drug: IVA
- Cohort C1: Triple Placebo (Placebo Comparator)
  Interventions: Drug: Matched Placebos
- Cohort C2 (Experimental)
  Interventions: Drug: VX-440; Drug: TEZ; Drug: IVA
- Cohort C2: Triple Placebo (Placebo Comparator)
  Interventions: Drug: Matched Placebos

INTERVENTIONS:
Drug: VX-440 — VX-440 was administered in TC with TEZ and IVA.
  Arms: Cohort C1; Cohort C2
Drug: TEZ — TEZ was administered as part of a fixed-dose combination (FDC) tablet (TEZ/IVA)
  Other Names: Tezacaftor; VX-661
  Arms: Cohort C1; Cohort C2
Drug: IVA — IVA was administered as part of a FDC tablet (TEZ/IVA) and as a mono tablet
  Other Names: Ivacaftor; VX-770
  Arms: Cohort C1; Cohort C2
Drug: Matched Placebos — Placebos matched to VX-440, TEZ, and IVA.
  Arms: Cohort C1: Triple Placebo; Cohort C2: Triple Placebo

SUMMARY:
This study evaluated the safety and pharmacokinetics of multiple ascending doses of VX-440 in combination with tezacaftor/ivacaftor (TEZ/IVA) (triple combination [TC]) administered for 13 days to healthy male and female subjects

ELIGIBILITY:
Inclusion Criteria:

* Female subjects of non-childbearing potential only.
* Body mass index (BMI) of 18.0 to 31.0 kg/m2, inclusive, and a total body weight >50 kg.
* Normal pulmonary function measurements, defined as forced expiratory volume in 1 second (FEV1) and forced vital capacity (FVC) both ≥80% of their predicted value at screening.

Exclusion Criteria:

* For female subjects: Pregnant or nursing subjects.
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency.
* History of hemolysis.
* Total bilirubin level >2 × ULN at Screening.

Other protocol defined Inclusion/Exclusion criteria applied.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2016-07-20 (Actual); Primary Completion 2016-09-14 (Actual); Study Completion 2016-09-14 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability were based on the number and assessment of adverse events (AEs) and serious adverse events (SAEs) | from baseline through safety follow-up visit (up to 29 days)

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) of VX-440, TEZ and its metabolites (M1-TEZ and M2-TEZ), and IVA and its metabolites (M1-IVA and M6-IVA) | from Day 1 through Day 18
Area under the concentration versus time curve during a dosing interval (AUCtau) of VX-440, TEZ and its metabolites (M1-TEZ and M2-TEZ), and IVA and its metabolites (M1-IVA and M6-IVA) | from Day 1 through Day 18
Observed pre-dose concentration (Ctrough) of VX-440, TEZ and its metabolites (M1-TEZ and M2-TEZ), and IVA and its metabolites (M1-IVA and M6-IVA) | from Day 1 through Day 18

CONTACTS AND LOCATIONS:
Locations (1):
- The Medicines Evaluation Unit, Manchester, United Kingdom